CLINICAL TRIAL: NCT06222515
Title: Novel Classification Algorism Derived From 3-day Bladder Diary for Female Storage Lower Urinary Tract Symptoms and Correlations of Clinical and Urodynamic Findings
Brief Title: Bladder Diary for Female Storage LUTS
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202303058RINC
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Urinary Urge Incontinence; Urinary Frequency More Than Once at Night; Stress Urinary Incontinence
Keywords: Storage; Lower urinary tract symptom; Female; Bladder diary
MeSH Terms: conditions — Urinary Incontinence, Urge; Nocturia; Urinary Incontinence, Stress; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with storage lower urinary tract symptom: The women with lower urinary tract symptoms, including urinary urgency (UU), stress urinary incontinence(SUI), urgency urinary incontinence (UUI), nocturia (N) and frequency (F).
  Interventions: Diagnostic Test: Bladder diary

INTERVENTIONS:
Diagnostic Test: Bladder diary — 3-day bladder diary record including fluid intake, urine amount, urgency and incontinence.

SUMMARY:
Storage urinary symptoms are the most complained of lower urinary tract symptoms (LUTS) and need further classification. This original study aims to derive a novel classification algorism for female storage LUTS according to a 3-day bladder diary (BD). Further feasibility of the application was also evaluated.

DETAILED DESCRIPTION:
Between July 2009 and December 2021, all women with storage lower urinary tract symptoms (LUTS) who visited the urogynecological department of a medical center were included. Women without complete data of a 3-day bladder diary (BD) were excluded from this study. The women were allocated into 12 groups according to the study flowchart based on their LUTS, including urinary urgency, stress urinary incontinence, urgency urinary incontinence, nocturia and frequency. MedCalc software was used for statistical analysis. Analysis of variance (ANOVA) was applied, and a P-value of less than 0.05 was considered as statistically significant. Post-hot analyses by the Student-Newman-Keuls test were performed only in those comparisons with p < 0.05 after ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Women more than 20-years-old
* With storage lower urinary tract symptoms
* Finished a 3-day bladder diary

Exclusion Criteria:

* No lower urinary tract symptoms
* Pregnant
* Incomplete data of bladder diary

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between July 2009 and December 2021, all women with storage LUTS who visited the urogynecological department of a medical center were included. Women without complete data of a BD were excluded from this study. The women were allocated into 12 groups according to the study flowchart based on their LUTS, including urinary urgency (UU), stress urinary incontinence(SUI), urgency urinary incontinence (UUI), nocturia (N) and frequency (F). MedCalc software was used for statistical analysis. Analysis of variance (ANOVA) was applied, and a P-value of less than 0.05 was considered as statistically significant. Post-hot analyses by the Student-Newman-Keuls test were performed only in those comparisons with p < 0.05 after ANOVA.
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Female lower urinary tract symptom classification | 3 days
  Classification of female lower urinary tract symptoms based on bladder diary, , including urinary urgency (UU), stress urinary incontinence(SUI), urgency urinary incontinence (UUI), nocturia (N) and frequency (F) and the combination of diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-chi Wu, MD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Pei-chi Wu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will be shared under reasonable request.

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Coyne KS, Wein AJ, Tubaro A, Sexton CC, Thompson CL, Kopp ZS, Aiyer LP. The burden of lower urinary tract symptoms: evaluating the effect of LUTS on health-related quality of life, anxiety and depression: EpiLUTS. BJU Int. 2009 Apr;103 Suppl 3:4-11. doi: 10.1111/j.1464-410X.2009.08371.x. PMID 19302497
- [Result] Hsiao SM, Lin HH. Medical treatment of female overactive bladder syndrome and treatment-related effects. J Formos Med Assoc. 2018 Oct;117(10):871-878. doi: 10.1016/j.jfma.2018.01.011. Epub 2018 Feb 15. PMID 29398096
- [Result] Hsiao SM, Su TC, Chen CH, Chang TC, Lin HH. Autonomic dysfunction and arterial stiffness in female overactive bladder patients and antimuscarinics related effects. Maturitas. 2014 Sep;79(1):65-9. doi: 10.1016/j.maturitas.2014.06.001. Epub 2014 Jun 20. PMID 25022469
- [Result] Hsiao SM, Liao SC, Chen CH, Chang TC, Lin HH. Psychometric assessment of female overactive bladder syndrome and antimuscarinics-related effects. Maturitas. 2014 Dec;79(4):428-34. doi: 10.1016/j.maturitas.2014.08.009. Epub 2014 Sep 3. PMID 25238744